CLINICAL TRIAL: NCT06165406
Title: Distal Radial Access for Diagnostic and Interventional Coronary Procedures in an All-comer Population: Observational Registry
Brief Title: Distal Radial Access for Coronary Procedures
Acronym: DISTAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Arnau de Vilanova (Other)
Collaborators: Hospital Universitario Torrecárdenas (Other); Hospital Regional de Malaga (Other); Hospital Universitari de Bellvitge (Other); Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Kristian Rivera, Principal Investigator, Hospital Arnau de Vilanova
Other Study IDs: CEIC-2804
Record Dates: First submitted 2023-11-28; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Vascular Access Complication; Coronary Artery Disease; STEMI; Non STEMI; Angina, Unstable; Angina, Stable; Artery Occlusion; Hematoma; Procedural Pain; Procedural Blood Vessel Puncture
Keywords: distal radial access; coronary procedures; ultrasound guided punction; vascular access; access-related complications; transradial access
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Angina, Stable; Arterial Occlusive Diseases; Hematoma; Pain, Procedural | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Distal radial access — Distal radial access for coronary procedures
  Other Names: coronary angiography; percutaneous coronary intervention; ultrasound-guided access

SUMMARY:
Distal radial access (DRA) in the anatomical snuffbox (AS) is a relatively novel approach that can be considered an alternative to trans radial access (TRA) for coronary procedures. Several observational and randomized studies have established its feasibility and safety, with evidence of certain advantages over TRA, such as a reduction in hemostasis time, a lower incidence of complications at the puncture site, and a lower incidence of radial artery occlusion (RAO). Notwithstanding that a recent randomized study reported a similar RAO rate between DRA and TRA, several meta-analyzes confirm the advantages of DRA, despite a consistently higher crossover rate.

The objective of this observational study is to assess the performance of the procedure and to compare clinical characteristics in an all-comer population undergoing diagnostic or interventional coronary procedures.

The main questions it aims to answer are:

* Determine the success rate of DRA and measure the incidence of RAO in an all-comer population undergoing coronary procedures.
* Compare the clinical and anatomical characteristics of patients with DRA for coronary procedures and determine predictors of failure of access.

DETAILED DESCRIPTION:
Introduction In recent decades, trans radial access (TRA) through the proximal radial artery has become the standard access site for performing diagnostic and therapeutic coronary procedures, its advantages over trans femoral access being demonstrated through multiple studies. such as reduction in access site complications and even reduction in mortality, especially in higher-risk patients.

There are circumstances in which anatomical variants can limit the clinical benefits of TRA, generating complications such as radial artery occlusion (RAO), which is by far the most frequent complication of this access, with a higher incidence at 24 h and recanalization after 30 days in 50% of patients. The presence of RAO limits access to future procedures, if necessary. The incidence of RAO reported in experienced centers remains high.

Distal Radial Access (DRA) through the anatomical snuffbox of the hand is a technique that has emerged in recent years and has been consolidated in multiple multicenter studies and meta-analyses to obtain arterial access in patients undergoing coronary angiography. and coronary intervention, which reduces the incidence of RAO, in addition to reducing hemostasis times, favoring patient and operator comfort compared to TRA.

DRA requires a slightly higher learning curve than TRA due to certain anatomical characteristics, such as the size of the distal radial artery, its depth, the presence of tortuosities, and the specific anatomical structures surrounding it. The DRA technique initially described was based on anatomical references (conventional puncture), however, the introduction of ultrasound as a puncture tool allows the operator to identify the size and course of the artery, in addition to a better assessment of the anatomy of the artery. area, thus avoiding injuries to them.

Most of the registries and clinical trials conducted to date are single centers, so the conduct of collaborative studies is of interest to determine the usefulness of different types of arterial access in coronary procedures.

OBJECTIVES Compare the clinical and procedural characteristics of patients undergoing diagnostic or therapeutic coronary procedures using DRA.

PRIMARY OBJECTIVE

1. Determine the success rate of DRA and measure the incidence of RAO.

SECONDARY OBJECTIVES

1. Compare the clinical (such as sex, age, weight, etc.) and anatomical characteristics (size of the proximal and distal radial artery size, depth of the distal radial artery) of patients with DRA.
2. Compare the time spent obtaining arterial access using DRA.
3. Assess the characteristics of the DRA procedure.
4. Assess the usefulness of ultrasound evaluation of the radial artery prior to DRA and US-guided DRA.
5. Investigate the predictors of failure for DRA.
6. Calculate the incidence of local complications related to DRA, radial spasm, puncture site hematoma, RAO, and presence of pseudoaneurysm of the radial artery.
7. Assess the operator's and patient comfort based on access.

STUDY DESIGN Prospective cohort of patients undergoing diagnostic or therapeutic coronary intervention, performed at the University Hospital Arnau de Vilanova in Lleida and open to other centers.

ELIGIBILITY:
Inclusion criteria:

* Patients who have undergone diagnostic or therapeutic coronary procedures using DRA in any clinical setting.
* Patients over 18 years of age.
* Presence of distal radial pulse.
* The Barbeau test was recommended but not mandatory.

Exclusion criteria:

* Previously known allergy to iodinated contrast and inability to receive premedication.
* Absence of distal radial pulse and distal radial artery not feasible by ultrasound.
* Women with the possibility of being pregnant.
* Inclusion in other clinical trials or registries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients who underwent diagnostic and therapeutic coronary procedures in an all-comer population using DRA between August 2020 and December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular access success | During the vascular access procedure.
  Defined when the introducer sheath can be placed appropriately through the punctured artery.

SECONDARY OUTCOMES:
Distal radial access time | During the vascular access procedure
  Begins when the anesthesia needle contacts the skin and ends when the introducer sheath has been properly placed.
Radial artery spasm | Throughout the procedure
  When at least two of the following five signs were met or only one of them after administration of a second dose of the spasmolytic agent, depending on the operator: persistent pain in the forearm, painful response to manipulation of the catheter, painful response to sheath withdrawal, difficulty in catheter manipulation after being trapped by the radial artery with considerable resistance to sheath withdrawal.
Total procedure time | Throughout the procedure
  Was considered from the moment the patient entered the catheterization laboratory until the patient left the catheterization laboratory.
Patient comfort during vascular access. | Throughout the procedure
  It was evaluated using a visual analog pain scale. It allows for measuring the intensity of the pain described by the patient. It consists of a horizontal line of 10 cm. On the left is the absence or lesser intensity, and on the right is the greatest intensity. The assessment will be mild pain if the patient rates the pain as less than 3, moderate pain if the rating is between 4 and 7, and severe pain if the rating is equal to or greater than 8.
Exposure to ionizing radiation | At the end of the procedure (up to 5 minutes).
  Was assessed using the dose area product (DAP) in Gy.m2
Access-related complications | At the end of the procedure (up to 6 hours).
  In-hospital radial artery occlusion was defined as the absence of anterograde flow signal on Doppler color ultrasound (US) distal to the radial artery 1-4 hours after the procedure was completed.
  The forearm hematoma related to DRA was defined according to the classification "Early discharge after transradial stimulation of the coronary arteries study" (EASY): grade I, <5cm in diameter; grade II, 5-10 cm in diameter; grade III, >10cm but distal to the elbow; grade IV that extends above the elbow; and grade V, anywhere with an ischemic threat to the hand.
  Radial artery dissection, pseudoaneurysms, and arteriovenous fistula were also considered vascular complications related to access.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Rivera, MD, Principal Investigator — University Hospital Arnau de Vilanova, Lleida Spain.
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Yes
After anonymization, all data collected during the study could be shared. Data obtained through this study may be provided to qualified researchers with academic interest in cardiovascular diseases. The approval of the request and the execution of all applicable agreements are prerequisites for the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data will be available from the publication of the study until 2 years later.
Access Criteria: The data will be shared with people interested in distal radial access through the contact email.